CLINICAL TRIAL: NCT03307343
Title: Effect of Reducing Sedentary Behavior on Blood Pressure
Acronym: RESET-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bethany Barone Gibbs, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19030297; R01HL134809 (NIH)
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Prehypertension
Keywords: sedentary behavior; light intensity physical activity; behavioral intervention; office workers; blood pressure; pulse wave velocity; randomized clinical trial
MeSH Terms: conditions — Hypertension; Prehypertension; Sedentary Behavior | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the participant group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will use behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts to target a 2-4 hour/day reduction in sedentary behavior.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Participants randomized to the control condition will receive no intervention during the study. After the 3-month assessment, control participants will be provided with a wrist-worn activity monitor and will be offered the 3-month delayed intervention if desired to aid in retention and recruitment.

INTERVENTIONS:
Behavioral: Intervention — The intervention will be delivered by trained research staff who are exercise physiologists or behavioral lifestyle counselors. This target reflects a recent expert statement concluding that desk-based workers should reduce workday sedentary behavior by 2-4 hr (by increasing standing and movement). The approach will combine: behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts. The initial in-person session will occur at the participant's office location. During months 2 and 3, one-on-one in-person meetings will occur at the research lab. Telephone intervention contacts will occur in the 3rd week of months 1-3.
  Other Names: Sedentary Behavior Reduction
  Arms: Intervention

SUMMARY:
This is a 2-arm, 3-month randomized trial comparing a novel sedentary behavior intervention vs. control in working adults (n=271). The primary outcome is resting systolic blood pressure (SBP) at 3 months; secondary outcomes will be resting diastolic blood pressure (DBP), ambulatory blood pressure (ABP), and carotid-femoral pulse wave velocity (cfPWV). Also, best practice objective activity monitoring will be leveraged in the analysis of ABP to account for recent activity and posture and will inform adherence and dose-response relationships.We will also measure plasma renin activity and aldosterone as a potential mechanism of blood pressure reduction, and insulin and glucose as exploratory outcomes.

DETAILED DESCRIPTION:
Hypertension (HTN) is the most common major risk factor for cardiovascular disease (CVD), affecting 1 in 3 American adults. Also, nearly another 1 in 3 adults has prehypertension (preHTN). Moderate-to-vigorous intensity physical activity (MVPA) is known to decrease BP. Guidelines recommend 150 min/week of MVPA performed in continuous bouts of ≥10 min (i.e., bouted MVPA). Sedentary behavior (SED), defined as sitting or reclining with low energy expenditure, has gained attention as a highly prevalent and distinct behavior from MVPA that is independently associated with higher BP, arterial stiffness, CVD, and mortality. These data, coupled with the fact that Americans spend more than half of the waking day in SED, suggest SED as a novel intervention target. Yet, despite heightened public perception of SED as a health risk, there is a dearth of randomized clinical trials demonstrating that SED reduction will lead to health benefits, including reduced BP. Decreasing SED more substantially could improve BP, but this remains unclear in the absence of larger randomized trials with effective SED interventions.

Thus, to test initial efficacy, the Effect of Reducing Sedentary Behavior on Blood Pressure (RESET-BP) has the following specific aims:

Specific aim 1: To evaluate the efficacy of our intervention targeting decreased sedentary behavior (SED) over 3 months. Outcomes include SBP (primary), DBP, ABP (nocturnal, daytime seated, daytime non-seated), and cfPWV. We hypothesize that the 3-month SED intervention will decrease SBP, DBP, ABP and cfPWV vs. controls

Specific Aim 2: To explore whether renin-angiotensin-aldosterone (RAAS) activation (increased plasma renin activity (PRA) and aldosterone) mediates changes in BP elicited by SED reduction

Specific Aim 3: To examine associations between achieved reductions in SED, increases in replacement behaviors (i.e., standing, other light-intensity physical activity (LPA), and BP reduction

These aims will be evaluated with a 2-arm, 3-month randomized trial comparing a novel SED intervention vs. control in 271 adults. The study will recruit adults with untreated, elevated blood pressure (SBP 120-159 mmHg or DBP 80-99 mmHg) and desk jobs that require prolonged SED to maximize the opportunity for SED reduction. The intervention will target currently recommended levels of SED reduction for desk-based employees (2-4 hours/day with frequent postural changes) and will use a behavioral intervention including individual in-person (1/month) and phone counselling (1/month) focused on goal setting, overcoming barriers, self-monitoring, social support, and stimulus control. In addition, the intervention will include environmental modification via provision of a sit-stand desk attachment and external prompting via text messaging and a wrist-worn inactivity prompter.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years
2. SBP 120-159 mmHg or DBP of 80-99
3. Inactive (Engages in less than 150 min/wk of moderate + 2 x vigorous intensity physical activity)
4. Currently perform deskwork for ≥ 20 hr/week at a desk compatible with the sit-stand attachment
5. Employment within an approximate 25-mile radius of the University of Pittsburgh
6. Stable employment (≥ 3 months in current job, plan to be in current job for the next 3 months)
7. Supervisor approval to join the intervention
8. Possession of a cellular phone able to receive text messages

Exclusion Criteria:

1. SBP ≥ 160 mmHg, DBP ≥ 100 mmHg
2. Use of antihypertensive or glucose controlling medication
3. Comorbid condition that would limit ability to reduce sedentary behavior (e.g. musculoskeletal condition, current chemotherapy)
4. History of ischemic heart disease, chronic heart failure, stroke, or chronic kidney disease
5. Unable to obtain consent from primary care provider or physician to participate
6. Current use of sit-stand/standing desk, sedentary behavior prompting device, enrollment in a weight loss or exercise study or program, recent (< 1 year) or planned bariatric surgery
7. Currently pregnant or pregnant in that last 6 months; breastfeeding currently or in the last 3 months
8. Plans to be away from your desk for an extended period (>1 week) during the study period

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Barone Gibbs, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Physical Activity and Weight Management Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the deidentified individual participant data collected during the trial will be shared (including the data dictionary).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication with no planned end date.
Access Criteria: Data access will be provided to researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Holmes AJ, Kline CE, Davis KK, Gordon BD, Stoner L, Quinn TD, Paley JL, Gibbs BB. Comparison of 24-Hour Movement Behaviors in Desk Workers Across Office and Work From Home Locations. J Occup Environ Med. 2025 Jul 1;67(7):e469-e477. doi: 10.1097/JOM.0000000000003380. Epub 2025 Mar 4. PMID 40165467
- [Derived] Quinn TD, Perera S, Conroy MB, Jakicic JM, Muldoon MF, Huber KA, Alansare AB, Holmes AJ, Barone Gibbs B. Impact of sedentary behaviour reduction on desk-worker workplace satisfaction, productivity, mood and health-related quality of life: a randomised trial. Occup Environ Med. 2025 Apr 16;82(2):61-68. doi: 10.1136/oemed-2024-109868. PMID 40011044
- [Derived] Barone Gibbs B, Perera S, Huber KA, Paley JL, Conroy MB, Jakicic JM, Muldoon MF. Effects of Sedentary Behavior Reduction on Blood Pressure in Desk Workers: Results From the RESET-BP Randomized Clinical Trial. Circulation. 2024 Oct 29;150(18):1416-1427. doi: 10.1161/CIRCULATIONAHA.123.068564. Epub 2024 Aug 21. PMID 39166323
- [Derived] Alansare AB, Paley JL, Quinn TD, Gibbs BB. Paradoxical Associations of Occupational and Nonoccupational Sedentary Behavior With Cardiovascular Disease Risk Measures in Desk Workers. J Occup Environ Med. 2023 Jul 1;65(7):e506-e513. doi: 10.1097/JOM.0000000000002873. Epub 2023 Apr 30. PMID 37130827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the vicinity of Pittsburgh, Pennsylvania using a variety of methods (physician's lists, research registries, university automated email blasts, etc.) between November 2017 and November 2022. The first participant was enrolled on January 3, 2018, and the last participant to complete data collection was on November 22, 2022.
Pre-assignment Details: 271 participants met inclusion criteria and were randomized to either the Sedentary Behavior Reduction Group or the No Contact Control Group. The majority of enrolled participants were excluded due to out of range blood pressure measurements and loss of interest.
Groups:
- Sedentary Behavior Intervention: The intervention will use behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts to target a 2-4 hour/day reduction in sedentary behavior.
- No Contact Control: Participants randomized to the control condition will receive no intervention during the study. After the 3-month assessment, control participants will be provided with a wrist-worn activity monitor and will be offered the 3-month delayed intervention if desired to aid in retention and recruitment.
Period: Overall Study
Arm/Group | Sedentary Behavior Intervention | No Contact Control
Started | 136 | 135
Completed | 134 | 129
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Pregnancy | 0 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention: The intervention will use behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts to target a 2-4 hour/day reduction in sedentary behavior.
  Intervention: The intervention will be delivered by trained research staff who are exercise physiologists or behavioral lifestyle counselors. This target reflects a recent expert statement concluding that desk-based workers should reduce workday sedentary behavior by 2-4 hr (by increasing standing and movement). The approach will combine: behavioral strategies (self-monitoring, goal setting, problem solving, social support, stimulus control), environment modification (sit-stand attachment), and proximal (activity prompter) and distal (text messages) external prompts. Face-to-face intervention lessons occurred in months 1, 2, and 3. Telephone intervention contacts will occur in the 3rd week of months 1-3.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 136 | 135 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.4) | 43.2 (11.5) | 45.2 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 82 | 163
  Male | 55 | 53 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 130 | 130 | 260
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 12 | 21
  White | 114 | 112 | 226
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Resting Systolic Blood Pressure
Description: Resting systolic blood pressure will be measured at baseline and follow-up using an oscillometric device after a 10-minute rest on two occasions
Time Frame: Baseline and Follow-Up (3 months)
Population: Systolic Blood Pressure (SBP)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sedentary Behavior Intervention | No Contact Control
Number analyzed (Participants) | 136 | 135
mm Hg
  Baseline Systolic Resting Blood Pressure | 129.5 (8.3) | 127.9 (9.2)
  Follow-Up Systolic Resting Blood Pressure | 124.3 (8.9) | 123.6 (10.9)

2. Secondary Outcome: Resting Diastolic Blood Pressure
Description: Resting diastolic blood pressure will be measured at baseline and follow-up using an oscillometric device after a 10-min rest on two occasions
Time Frame: Baseline and Follow-Up (3 months)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sedentary Behavior Intervention | No Contact Control
Number analyzed (Participants) | 136 | 135
mm Hg
  Resting Baseline Diastolic Blood Pressure | 82.7 (7.0) | 82.9 (6.4)
  Resting Follow-Up Diastolic Blood Pressure | 79.7 (7.8) | 79.9 (6.9)

3. Secondary Outcome: 24-Hour Systolic/Diastolic Ambulatory Blood Pressure
Description: Ambulatory blood pressure will be measured at baseline and 3-month follow-up during a workday and overnight (24 hours total) at the beginning and end of the study
Time Frame: Baseline and Follow-Up (3 months)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sedentary Behavior Intervention | No Contact Control
Number analyzed (Participants) | 136 | 135
mm Hg
  24-Hour Baseline Systolic Blood Pressure | 130.2 (8.8) | 129.5 (9.5)
  24-Hour Baseline Diastolic Blood Pressure | 78.1 (6.4) | 78.4 (6.4)
  24-Hour Follow-Up Systolic Blood Pressure | 130.2 (10.4) | 129.7 (9.8)
  24-Hour Follow-Up Diastolic Blood Pressure | 78.6 (7.5) | 77.9 (6.9)

4. Secondary Outcome: Pulse Wave Velocity
Description: Carotid-femoral and carotid-radial pulse wave velocity will be measured at baseline and follow-up following a 10-min supine rest via tonometry.
Time Frame: Baseline and Follow-Up (3 months)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Intervention | Control
Number analyzed (Participants) | 136 | 135
m/s
  Baseline carotid-femoral | 8.22 (1.70) | 7.66 (1.20)
  Baseline carotid-radial | 9.09 (1.30) | 8.97 (1.05)
  Follow-up carotid-femoral | 8.29 (1.76) | 7.68 (1.18)
  Follow-up carotid-radial | 9.16 (1.23) | 9.07 (1.11)

5. Secondary Outcome: Plasma Renin Activity
Description: Plasma Renin Activity (PRA) will be measured at baseline and 3 month follow-up.
Time Frame: Baseline and Follow-Up (3 months)
Population: Participants who had both baseline and follow-up valid blood samples were included. Change descriptive results are reported.
Measure: Mean (Standard Deviation); unit: ng/mL/hr
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 85
ng/mL/hr | -0.16 (1.02) | 0.07 (0.75)

6. Secondary Outcome: Aldosterone
Description: Aldosterone will be measured at baseline and 3 month follow-up.
Time Frame: Baseline and Follow-Up (3 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 87 | 86
ng/dL | -0.52 (49.25) | 13.14 (45.88)

7. Other Pre Specified Outcome: Glucose
Description: Glucose will be measure at baseline and 3 month follow-up.
Time Frame: Baseline and Follow-up (3 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 93
mg/dL | -2.81 (13.83) | 0.76 (12.00)

8. Other Pre Specified Outcome: Insulin
Description: Insulin will be measured at baseline and 3 month follow-up.
Time Frame: Baseline and Follow-Up (3 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 95 | 93
U/mL | -1.44 (15.39) | -0.02 (6.11)

9. Other Pre Specified Outcome: Weight
Description: Weight will be measured by digital scale at baseline and 3 month follow-up.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 136 | 135
kg
  Baseline Weight | 88.1 (18.9) | 90.8 (22.4)
  Follow-up Weight | 87.9 (18.6) | 91.2 (21.9)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were assessed prospectively at each research interaction and systematically at 3-month follow-up.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/135
Serious Adverse Events (participants affected / at risk) | 4/136 | 4/135
Other Adverse Events (participants affected / at risk) | 32/136 | 24/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=136) | Control (N=135)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hospitalization due to diabetes (Endocrine disorders) | 1 (1) | 0 (0)
Grand Mal Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=136) | Control (N=135)
Bruising on Arm from ABPM (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Arm Pain and Redness from ABPM Cuff (Injury, poisoning and procedural complications) | 4 (4) | 4 (5)
Petechiae from ABPM Measurement (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin Irritation from Monitor Wear (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)
Vasovagal Reaction Following Blood Draw (General disorders) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Positive COVID-19 Diagnosis (Infections and infestations) | 2 (2) | 1 (1)
Concussion from Object Falling on Head (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Started taking disallowed medication (Metformin) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back, Joint, Arthritis Pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (6)
Eating Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Planned Surgical Procedures (Surgical and medical procedures) | 1 (1) | 2 (2)
Diabetes Diagnosis (Endocrine disorders) | 1 (1) | 0 (0)
Diverticulitis Event/Diagnosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergic Reaction (difficulty breathing) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Falls and Accidents (Injury, poisoning and procedural complications) | 6 (8) | 0 (0)
Muscle/Tendon Injuries (Injury, poisoning and procedural complications) | 4 (7) | 0 (0)
Traumatic Incident (Social circumstances) | 1 (1) | 0 (0)
Tick Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT03307343/Prot_SAP_000.pdf